CLINICAL TRIAL: NCT03850340
Title: Retrospective Evaluation of the Review of Automated Ventilator Data's Effect on the Incidence of Ventilator Associated Events in a Medical Surgical Intensive Care Unit
Brief Title: Evaluation of the Review of Automated Ventilator Data's Effect on the Incidence of Ventilator Associated Events in a Medical Surgical Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's/Candler Health System (Other)
Responsible Party: Principal Investigator, Harold Julius-Augustus Oglesby, Manager, Pulmonary Medicine, St. Joseph's/Candler Health System
Other Study IDs: IRB# 18-027
Record Dates: First submitted 2019-01-29; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Ventilator Associated Events
Keywords: Ventilator Associated Conditions; Infection Related Ventilator Associated Conditions; Probable Ventilator Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be a retrospective, observational analysis study of ventilator patients in the Medical Surgical Intensive Care unit being monitored via automated near real-time ventilator analytical software.

DETAILED DESCRIPTION:
This study will be a retrospective review of data via chart review of all mechanically ventilated patients in an Intensive Care unit meeting our inclusion criteria during the pre-implementation and post-implementation phases of the study. Data will be collected and a detailed analysis of outcomes will be performed. The major parameters that will be measured will focus on the rate of ventilator associated events during each phases of the analysis.

Ventilator associated events will be defined as Ventilator associated Conditions (VACs), Infection related Ventilator Associated Conditions (IVACs) and Probable Ventilator Associated Pneumonias (PVAPs). According to the Center for Disease & Control a VAC occurs after a patients has ≥ 2 days of stable or decreasing minimum FiO2 or PEEP values and then experiences at least one of the following: increased in the daily minimum FiO2 of ≥ 0.20 over the daily minimum FiO2 in the baseline period, sustained for ≥ 2 calendar days or increase in the daily minimum PEEP values of ≥ 3 cmH2O over the daily minimum PEEP in the baseline period sustained for ≥ 2 calendar days. An IVAC is defined as the occurrence on or after calendar day 3 of mechanical ventilation and within 2 calendar days before or after the onset of worsening oxygenation, the patient meets both of the following criteria: 1) Temperature > 38C, or white blood cell count ≥ 12,000 cells/mm3 or ≤ 4,000 cells/mm3 and a new antimicrobial agents(s) is started for ≥ 4 calendar days. A PVAP is occurs when a patient meets the criteria for a VAC and IVAC and one of the following criteria are met: 1) Purulent respiratory secretions (from one or more specimen collections). 2) Positive culture (qualitative, semi-quantitative) of sputum, endotracheal aspirate, bronchoalveolar lavage, lung tissue, or protected specimen brushing.

ELIGIBILITY:
Inclusion Criteria:

* includes all mechanically ventilated patients in the Intensive Care Unit above the age of 18 years of age and who were mechanically ventilated for ≥ 3 days.

Exclusion Criteria:

* any patients under the age of 18 or mechanically ventilated for < 3days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: includes all mechanically ventilated patients in the study center's Medical-Surgical Intensive Care Unit above the age of 18 years of age and who were mechanically ventilated for ≥ 3 days.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-31 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ventilator Associated Events | 03/01/2014 until 02/28/2019
  Measure of the number of occurrences of ventilator associated events